CLINICAL TRIAL: NCT04349748
Title: The Effect of Providing mHealth Intervention of Partner Notification to Protect MSM From HIV and Sexually Transmitted Diseases Infection: a Pragmatic Stepped Wedge Cluster Randomized Controlled Trial
Brief Title: MHealth Intervention of HIV and STDs Partner Notification for MSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute on Drug Dependence, China (Other)
Collaborators: Man Wellness Center, Beijing, China (Unknown)
Responsible Party: Principal Investigator, ZhongweiJia, Professor, Director of Center for Drug Abuse Control and Prevention, National Institute on Drug Dependence, China
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NIDD-HIV
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: HIV/AIDS; Sexually Transmitted Diseases; Prevention
Keywords: HIV/AIDS; sexually transmitted disease (STD); men who have sex with men (MSM); partner notification; mHealth application; stepped wedge cluster randomized controlled trial
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Homosexuality | interventions — Contact Tracing

STUDY DESIGN:
Intervention Model Description: This study is not a conventional crossover design,we use a pragmatic stepped-wedge cluster-randomised design.The study lasts for 2.5 years, which is divided to five continuous observation periods (every six months).The sixteen districts are assigned to four arms randomly.Four arms began recruiting participants at the same time,and at the first observation period,all groups were given health education and regular HIV and STDs testing prompting service,the two services above are given continuously for five observation periods.At the second observation period,the first group is given permission to query health status (partner notification) through app,but the other three groups do not.At every observation period after that (the third to fifth observation period),the three groups will be given permission to query health status one by one.Once a group is given the permission,it is retained until the end of study.
Who Masked: Outcomes Assessor
Masking Description: Because partner notification is a kind of behavioral intervention, participants know what intervention they receive. However, we take efforts to reduce the bias caused by the non-blind design. At the beginning of the research, participants, care providers, and researchers who participate in participants management will not know the randomized scheme. The partner notification will be opened to participants sequentially by the predetermined computer program, and does not need care providers and researchers to implement the intervention manually. The care providers and researchers do not know the implementation of partner notification unless the participants tell them whether they can use the function on their own initiative. Even the care providers know that, the operation and results of the HIV and STDs testing will not be affected. At last, the outcomes assessors do not know the randomized scheme in data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): The group is given health education, regular HIV and STDs testing prompting service in the whole study, and permission to query health status (partner notification) through app from the second observation period. HIV and STDs testing and questionnaire are given to the participants when they receive the testing service.
  Interventions: Behavioral: Health education, and regular HIV and STDs testing prompting service; Behavioral: Health status inquiry through app (partner notification)
- Group 2 (Experimental): The group is given health education, regular HIV and STDs testing prompting service in the whole study, and permission to query health status (partner notification) through app from the third observation period. HIV and STDs testing and questionnaire are given to the participants when they receive the testing service.
  Interventions: Behavioral: Health education, and regular HIV and STDs testing prompting service; Behavioral: Health status inquiry through app (partner notification)
- Group 3 (Experimental): The group is given health education, regular HIV and STDs testing prompting service in the whole study, and permission to query health status (partner notification) through app from the fourth observation period. HIV and STDs testing and questionnaire are given to the participants when they receive the testing service.
  Interventions: Behavioral: Health education, and regular HIV and STDs testing prompting service; Behavioral: Health status inquiry through app (partner notification)
- Group 4 (Experimental): The group is given health education, regular HIV and STDs testing prompting service in the whole study, and permission to query health status (partner notification) through app from the fifth observation period. HIV and STDs testing and questionnaire are given to the participants when they receive the testing service.
  Interventions: Behavioral: Health education, and regular HIV and STDs testing prompting service; Behavioral: Health status inquiry through app (partner notification)

INTERVENTIONS:
Behavioral: Health education, and regular HIV and STDs testing prompting service — Health education through app for once a week, and regular HIV and STDs testing prompting service (every month through app) are given to the participants at the beginning of the study and last for the whole five observation periods.
Behavioral: Health status inquiry through app (partner notification) — The permission to query health status through app (partner notification) is given to participants (participants can query their potential sexual partner's status of HIV, syphilis, hepatitis B, and hepatitis C respectively through app) at the specific observation period,and the permission is retained until the end of study.

SUMMARY:
Men who have sex with men (MSM) have become a focus of HIV and other sexually transmitted diseases (STD) control in China. Most of MSM who seek causal partners through online dating platforms do not know their sexual partners' real HIV and STDs infection status, which leads to more high risk status, especially for sexual behaviors. Effective Internet-based partner notification is urgently warranted to increase their risk awareness and prevent HIV and STDs transmission. This study developed an app which can help MSM to query recent HIV and other STDs statuses each other from the testing platform in order that they can find a relatively safety sexual partners and reduce risk of HIV infection.

DETAILED DESCRIPTION:
Because most of the recent "Partner Notification" methods are a kind of afterwards remedial measures and will fail to find some of the infected MSM, researchers propose a preventive measures before they meet together. For MSM who are seeking potential sexual partners through Internet, researchers will encourage them to query health status before they decide to meet each other in order to promote their healthy self-responsibility consciousnes including avoiding HIV and other STDs infection, which will form a real ,digital MSM cohort. Researchers designed a pragmatic stepped wedge cluster randomized controlled trial to evaluate the effect of an intervention paradigm that provides HIV, syphilis, hepatitis B, and hepatitis C status partner notification based on the existing HIV and STDs control methods through an mHealth application (app), to reduce HIV and STDs incidences among MSM in China. More than 6000 MSM of 16 districts in Beijing, China will be grouped into four arms, each arm will cover four indepednent districts of Beijing randomly. The four arms will be randomized to sequentially initiate partner notification intervention through the app at 6-month intervals. All participants will be provided informed consent in the app after a full explanation of the protocol design. Researchers expect that the HIV incidence will be significantly lower and the secondary outcomes will also be better after partner notification intervention. The feasible and affordable public health management paradigm will have implications for HIV and STDs prevention and control among MSM and other key populations.

ELIGIBILITY:
Inclusion criteria:

1. biologically male,
2. had oral or anal sex with men at least once during their lifetime,
3. 15 years of age or older,
4. had no difficulty using a mobile phone,
5. willing to provide their mobile phone numbers to serve as the unique identification numbers of the app's self-query and partner notification functions,
6. willing to use the app's function modules,
7. willing to complete the questionnaire for the research,
8. willing to continuously receive HIV and STDs testing and consulting services provided by the CBO our research setting at,
9. willing to complete the informed consent document.

Exclusion criteria:

1.had serious physical disabilities or mental diseases.

Min Age: 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6172 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
HIV positive seroconversion rate (HIV incidence) | through study completion, an average of six months
  The number of HIV positive seroconversions divided by the total number of person-years.
Additional cost of the intervention | through study completion, an average of six months
  The total cost and average cost for per participant of the integrated intervention model and each additional intervention/service based on the existing HIV prevention measures provided as before.

SECONDARY OUTCOMES:
Syphilis positive seroconversion rate (Syphilis incidence) | through study completion, an average of six months
  The number of syphilis seroconversions divided by the total number of person-years.
Hepatitis B positive seroconversion rate (Hepatitis B incidence) | through study completion, an average of six months
  The number of hepatitis B seroconversions divided by the total number of person-years.
Hepatitis C positive seroconversion rate (Hepatitis C incidence) | through study completion, an average of six months
  The number of hepatitis C seroconversions divided by the total number of person-years.
HIV and related diseases transmission among social networks | through study completion, an average of 1 year
  Based on the partner notification information, we will construct the transmission networks of HIV and other STDs (syphilis, hepatitis B, and hepatitis C) among participants, and analyze the characteristics of these networks and factors associated with transmission of these diseases.
Testing adherence | through study completion, an average of 1 year
  The proportion of participants whose every adjacent testing interval is no more than 3 months as recommended by China CDC.
Additional cost for finding per seroconversion | through study completion, an average of six months
  The total additional cost of the integrated intervention model based on the existing HIV prevention measures provided as before divided by the total number of the HIV and STDs seroconversions.
Frequency of utilization for each intervention/service | through study completion, an average of six months
  The total frequency and average frequency for per participant of utilization for each intervention/service, such as health education, partner notification, HIV and STDs testing and so on.
Satisfaction of the interventions and services | through study completion, an average of six months
  This indicator is measured by the follow-up questionnaires as the degree of satisfaction for participants of HIV and STDs testing service, health education, partner notification and other app's functions.
Knowledge of HIV and related STDs | through study completion, an average of six months
  This indicator is measured by the baseline and follow-up questionnaires, and we use the score of knowledge questions in the questionnaires to represent participants' level of knowledge.
Attitudes of HIV and STDs testing, safe sexual behaviors and partner notification | through study completion, an average of six months
  The attitudes are collected by these questions in the baseline and follow-up questionnaires.
Sexual behaviors | through study completion, an average of six months
  They are measured by questionnaires, including questions about the number of different kinds of sexual partners, frequency of anal sex, condom use, and partner notification implementation.
Substance use behaviors | through study completion, an average of six months
  This indicator is measured by questionnaires about participants' usage about methamphetamine, heroin, ecstasy, and some other sex-promoting drugs.
Psychological status | through study completion, an average of six months
  SAS (self-rating anxiety) scale and SDS (self-rating depression) scale are used to measure participants' psychological status through questionnaires. The higher scores of the two scares mean the worse outcomes.
Referral rate of HIV and related STDs | through study completion, an average of six months
  The proportion of new HIV and STDs infections who have received treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongwei Jia, Prof. PhD, Principal Investigator — National Institute on Drug Dependence, Peking University,China

IPD SHARING:
Plan to Share IPD: Yes
1. Study Protocol,part of study report and data will be published in journals;
  2. Researchers can contact the principal investigator(PI:ZhongweiJia) for IPD through email two years after the end of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Two years after the end of the trial
Access Criteria: Data applicants should send email to PI. Real personal basic information (name, unit, title, etc.), detailed description of required data (required variables,etc.), and research plan should be included in the email. Our team will discuss the research proposal and reply as soon as possible

REFERENCES:
- [Background] Brown LB, Miller WC, Kamanga G, Nyirenda N, Mmodzi P, Pettifor A, Dominik RC, Kaufman JS, Mapanje C, Martinson F, Cohen MS, Hoffman IF. HIV partner notification is effective and feasible in sub-Saharan Africa: opportunities for HIV treatment and prevention. J Acquir Immune Defic Syndr. 2011 Apr 15;56(5):437-42. doi: 10.1097/qai.0b013e318202bf7d. PMID 22046601
- [Background] Tsega A, Udeagu CC, Begier EM. A comparison of partner notification effectiveness in African-, Caribbean-, and United States-born HIV-infected Blacks in New York City. AIDS Patient Care STDS. 2012 Jul;26(7):406-10. doi: 10.1089/apc.2011.0313. Epub 2012 Jun 4. PMID 22663166
- [Background] Rosenberg NE, Mtande TK, Saidi F, Stanley C, Jere E, Paile L, Kumwenda K, Mofolo I, Ng'ambi W, Miller WC, Hoffman I, Hosseinipour M. Recruiting male partners for couple HIV testing and counselling in Malawi's option B+ programme: an unblinded randomised controlled trial. Lancet HIV. 2015 Nov;2(11):e483-91. doi: 10.1016/S2352-3018(15)00182-4. Epub 2015 Oct 22. PMID 26520928
- [Background] Yan X, Lu Z, Zhang B, Li Y, Tang W, Zhang L, Jia Z. Protecting Men Who Have Sex With Men From HIV Infection With an mHealth App for Partner Notification: Observational Study. JMIR Mhealth Uhealth. 2020 Feb 19;8(2):e14457. doi: 10.2196/14457. PMID 32130147
- [Derived] Yan X, Li Y, Su H, Xing Y, Zhang B, Lu Z, Jia Z. Protect MSM from HIV and other sexually transmitted diseases by providing mobile health services of partner notification: protocol for a pragmatic stepped wedge cluster randomized controlled trial. BMC Public Health. 2020 Jul 14;20(1):1107. doi: 10.1186/s12889-020-09162-x. PMID 32664934